CLINICAL TRIAL: NCT04861935
Title: Ultrasound Guided Investigation Of The Anatomical Features For Caudal Block In Children With Sacral Dimple
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Celal Kaya, Principal Investigator, MD, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 72109855-604.01.01-231115
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Sacrococcygeal Disorder
Keywords: pediatric, sacral dimple, ultrasound

STUDY DESIGN:
Intervention Model Description: Two groups were formed as those with and without dimples in the sacral region.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound evaluation of sacral region in normal pediatric patients (Placebo Comparator): Ultrasound evaluation of sacral region will be performed to detect spinal abnormality.
  Dural sac level and its distance to estmated injection site, optimal entry angle for caudal block will be measured.
  Interventions: Device: ultrasound evaluation
- ultrasound evaluation of sacral region in patients with sacral dimple (Active Comparator): Ultrasound evaluation of sacral region will be performed to detect spinal abnormality.
  Dural sac level and its distance to estmated injection site, optimal entry angle for caudal block will be measured.
  Interventions: Device: ultrasound evaluation

INTERVENTIONS:
Device: ultrasound evaluation — ultrasound evaluation of normal patients and patients who have a sacral dimple

SUMMARY:
When dimples are detected in the sacral region, most practitioners consider it to be a sign of spinal anomaly and avoid caudal block. Ultrasound guided investigation of the anatomical features for caudal block in normal children and in children with sacral dimple will be informative for practitioners.

DETAILED DESCRIPTION:
A dimple over the sacrum may be an isolated finding or a sign of underlying spinal abnormality. Therefore, most practitioners are confused to perform a caudal block. Ultrasonography is a safe and cost effective screening tool in pediatric patients. Ultrasound guided investigation of the anatomical features of sacral region may play a key role to eliminate suspicions. It is possible to detect spinal abnormalities and also measuring dural sac level, distance between dural sac and estimated needle insertion site or needle entry angle. In this study, we will examine whether there is a difference between normal children and children with dimple in the sacral region.

ELIGIBILITY:
Inclusion Criteria:

-Children aged 1-72 months who are taken to the operating room for any reason

Exclusion Criteria: Patients with

* spinal anomalies,
* history of prematurity,
* neurological disorder
* syndromic illness.

Ages: 1 Month to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
ultrasound measurement-1 | 1 min
  Dural sac level (mm)
ultrasound measurement-2 | 1 min
  distance between injection site and dural sac(mm)
ultrasound measurement-3 | 1 min
  optimal entry angle (0-angle degree) for caudal block

SECONDARY OUTCOMES:
ultrasound evaluation of sacral region | 10 minutes
  searching for spinal abnormalites in patients with sacral dimple

CONTACTS AND LOCATIONS:
Overall Officials: Guner Kaya, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Schwartz D, Al-Najjar H, Connelly NR. Caudal block in a child with a sacral dimple utilizing ultrasonography. Paediatr Anaesth. 2011 Oct;21(10):1073-4. doi: 10.1111/j.1460-9592.2011.03621.x. No abstract available. PMID 21981093
- [Background] Choi JH, Lee T, Kwon HH, You SK, Kang JW. Outcome of ultrasonographic imaging in infants with sacral dimple. Korean J Pediatr. 2018 Jun;61(6):194-199. doi: 10.3345/kjp.2018.61.6.194. Epub 2018 Jun 25. PMID 29963103